CLINICAL TRIAL: NCT05224791
Title: A Retrospective Multicenter Comparison of Laparoscopic and Robotic-Assisted Roux-en-Y Gastric Bypass and Sleeve Gastrectomy
Brief Title: A Retrospective Multicenter Comparison of Laparoscopic and Robotic-Assisted Roux-en-Y Gastrectomy
Status: Recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Collaborators: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: 015.WMP.2020.D
Record Dates: First submitted 2020-11-11; First posted 2022-02-04 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Laparoscopic Sleeve Gastrectomy; Sleeve Gastrectomy
Keywords: Sleeve Gastrectomy; laparoscopic; robotic-assisted RYGB
MeSH Terms: interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastric Bypass: The RYGB connects a limb of the intestine to a much smaller stomach pouch, which prevents the bile from entering the upper part of the stomach and esophagus, thereby effectively bypassing the remaining stomach and first segment of the small intestine.
  Interventions: Procedure: Roux-en-Y Gastric Bypass; Procedure: Sleeve Gastrectomy
- Sleeve Gastrectomy: The SG is a restrictive procedure in which a partial left gastrectomy of the fundus and body of the stomach is performed in order to create a long tubular "sleeve" along the lesser curvature. The weight loss and resolution of comorbidities are attributed not only to the restrictive nature of the procedure but also to restriction by the pylorus, decreased ghrelin, increased satiety, increased gastric emptying, and faster small bowel transit times with a component of malabsorption.
  Interventions: Procedure: Roux-en-Y Gastric Bypass; Procedure: Sleeve Gastrectomy

INTERVENTIONS:
Procedure: Roux-en-Y Gastric Bypass — The RYGB connects a limb of the intestine to a much smaller stomach pouch, which prevents the bile from entering the upper part of the stomach and esophagus, thereby effectively bypassing the remaining stomach and first segment of the small intestine.
  Other Names: RYGB
Procedure: Sleeve Gastrectomy — The SG is a restrictive procedure in which a partial left gastrectomy of the fundus and body of the stomach is performed in order to create a long tubular "sleeve" along the lesser curvature. The weight loss and resolution of comorbidities are attributed not only to the restrictive nature of the procedure but also to restriction by the pylorus, decreased ghrelin, increased satiety, increased gastric emptying, and faster small bowel transit times with a component of malabsorption
  Other Names: SG

SUMMARY:
The prevalence of obesity has tripled in the last 50 years with presently about 1.7 billion of the world population aged 18 years and over either overweight or obese.1 In the US alone, 35% of the population is obese.2 Although alternative surgical approaches are available, bariatric surgery results in substantial and durable weight reduction for the majority of patients, making it the most effective treatment for severe obesity.3 In the battle to reduce the invasiveness of bariatric procedures, laparoscopy has become the gold standard approach for virtually all bariatric surgery procedures in the years since it was first used for gastric bypass by Wittgrove and colleagues in 1993.5 Available data shows perioperative patient-oriented advantages of laparoscopy when compared with open surgery, including a shorter hospital stay, decreased postoperative pain, and enhanced postoperative recovery.6 The Agency for Healthcare Research and Quality (AHRQ) reported significant improvements in the safety of metabolic/bariatric surgery due in large part to improved surgical techniques.7 The risk of death is about 0.1%8 and the overall likelihood of major complications is about 4%.9 Performing bariatric surgery laproscopically can be demanding in many situations because of large livers and substantial visceral fat that limit the working space and make exposure, dissection, and reconstruction difficult.10 Similarly, thick abdominal walls may cause excessive torque on instruments. Under such situations, surgeons' ergonomics become a serious concern.11 Use of robotics in bariatric surgery has been evolving since Cadiere and colleagues reported the first case in 1999.12 Robotic surgery has provided the surgeons with the advantage of three-dimensional vision as well as increased dexterity and precision by downscaling surgeon's movements enabling a fine tissue dissection and filtering out physiological tremor.13 It overcomes the restraint of torque on ports from thick abdominal wall, and minimizes port site trauma by remote center technology.14 Although Roux-en-Y gastric bypass (RYGB) is considered by many to be the gold standard procedure for weight loss,4 several studies demonstrate that sleeve gastrectomy (SG) and RYGB provide comparable weight loss.15 In fact, utilization of SG significantly increased from 9.3% in 2010 to 58.2% in 2014.16

DETAILED DESCRIPTION:
Procedure Description 1.2.1 Roux-en-Y Gastric Bypass The RYGB connects a limb of the intestine to a much smaller stomach pouch, which prevents the bile from entering the upper part of the stomach and esophagus, thereby effectively bypassing the remaining stomach and first segment of the small intestine. 21 The first step of RYGB involves the creation of the gastric pouch. The angle of His is identified with the fundus retracted laterally. The peritoneum, over the angle of His, is dissected with ultrasonic shears or scissors and carried posterior to identify the path for a linear stapler and the left crus of the diaphragm. Next, the mesentery to the lesser curve of the stomach is divided by a stapler. Once the retrogastric plane in the lesser curve is created, two serial applications of stapler will be used to create a 20 mL gastric pouch. 21 The second step is the creation of jejunojejunostomy. A stapler is utilized to create the anastomosis. The common enterotomy is closed with either a single running layer of 2-0 Vicryl or a second firing stapler. Finally, the gastrojejunal anastomosis is created and the Roux limb is pulled up to the level of the gastric pouch. 21

1.2.2 Sleeve Gastrectomy The SG is a restrictive procedure in which a partial left gastrectomy of the fundus and body of the stomach is performed in order to create a long tubular "sleeve" along the lesser curvature. The weight loss and resolution of comorbidities are attributed not only to the restrictive nature of the procedure but also to restriction by the pylorus, decreased ghrelin, increased satiety, increased gastric emptying, and faster small bowel transit times with a component of malabsorption.17-20

1.2 Aim(s)/Objective(s) The overall aim of this study is to evaluate and compare outcomes associated with robotic-assisted and laparoscopic bariatric surgery.

1.3 Rationale for the Study Studies to date have drawn partial contrasting conclusions when comparing robotic-assisted and laparoscopic bariatric surgery. There is a need to collect more scientific evidence data around the clinical outcomes of bariatric surgery performed with either robotic-assisted or laparoscopic surgery to describe the potential advantages of these techniques.

1.4 Hypothesis 1.4.1 Primary Hypothesis We hypothesize that the RYGB will indicate better outcomes compared to the SG.

2. OBJECTIVES AND STUDY OUTCOME MEASURES 2.1. Study Objectives The primary objective of this study is to retrospectively compare perioperative outcomes through discharge and short-term outcomes through 30 days after robotic-assisted and laparoscopic bariatric surgery.

2.2. Study Outcome Measures Baseline patient characteristics, intraoperative, post-operative, and short-term clinical data will be obtained from hospital records for a total of up to approximately 400 robotic-assisted and laparoscopic cases among the four subgroups: robotic-assisted RYGB, robotic-assisted SG, laparoscopic RYGB, and laparoscopic SG.

3. STUDY DESIGN This is a multi-center, retrospective chart review study of all consecutive cases of RYGB and SG, performed by participating surgeons at their respective institutions that meet the study inclusion and exclusion criteria.

The chart review will be performed in a reverse chronological order starting at a minimum of 30 days prior to IRB approval of the study at the site until and going back to 2017 (i.e. most current cases in 2020 and chronologically going back through 2017). Study initiation at the participating site will occur once a research agreement has been executed between Intuitive Surgical and the participating institution/ investigator and after IRB approval has been obtained.

It is anticipated that the retrospective chart review will span the period between January 1, 2017 through 30 days prior to IRB approval of the study at each institution. Perioperative and short-term clinical data will be obtained from institutional records. Each participating site and the participating surgeons at those institutions will contribute approximately a minimum of 10 to a maximum of 50 cases to a subgroup. The chart review and data collection will be performed in a reverse chronological order starting at 30 days prior to IRB approval of the study at the institution to 2017.

All the data variables will be documented in the case report forms. This section will provide an overview of the data collected which will include, but are not limited to, the following:

* Pre-Operative Information: Demographics (e.g. age, gender), patient characteristics (e.g. BMI, ASA Class), and pre-operative medical history (e.g. tobacco use, previous abdominal surgery, comorbidities: hypertension, cardiopulmonary disease, diabetes)
* Intra-Operative Data: Operative time, total OR time, bariatric procedure (robotic-assisted RYGB or SG and Laparoscopic RYGB or SG), concomitant procedures, transfusions, conversions, intraoperative adverse events
* Post-Operative Data (up to discharge): Post-operative adverse events, discharge status, hospital length of stay, information on enhanced recovery program
* Short-Term Follow-Up Data (up to 30 days post-discharge): Adverse events up to 30 days, re- admissions, re-operations related to the index procedure Please refer to the case report forms for complete details of data to be collected. Information regarding adverse events will be collected through this study; a list of applicable adverse events can be found below.

Because the data will have been de-identified and is archival in nature, there will be no active subject recruitment and no patient consenting is required. A study specific Informed Consent Waiver for retrospective data collection will be obtained for this study, as required by the institution's IRB policy.

The study duration is anticipated to be approximately 18 months.

* The site activation consisting of IRB submission/approvals, contract execution, and training is anticipated to be completed in approximately 3 to 4 months
* Chart review, data collection, and entry are anticipated to be completed in approximately 6 to 8 months
* Data review is anticipated to be completed in approximately 2 months
* Data analysis is anticipated to be completed in approximately 4 months Study Training All investigators/ site personnel will be trained on the study protocol at a Site initiation visit or at another appropriate training session. Site initiation visit will be scheduled only upon receiving a fully executed data collection agreement and IRB approval. Training of investigators and site study personnel will include, but are not limited to, the investigational plan, protocol requirements, CRF completion, EDC training, recording of adverse events, and study personnel responsibilities related to study compliance and conduct.

Adverse Events Adverse event data will be collected only for those associated with the primary bariatric procedures (RYGB and SG procedures) requiring intervention.

The investigator will be responsible for reviewing all the adverse event case report forms. A detailed list of adverse events is provided in the case report forms. Some examples of commonly anticipated intraoperative and post-operative adverse events are provided below but reported adverse events are not limited to the following.

* Examples of intraoperative adverse events

  * Bleeding requiring an intervention
  * Visceral injury including but not limited to injury to liver, injury to diaphragm, injury to spleen
  * Vascular injury including major vascular injury requiring intervention
  * Adverse events related to anesthesia (prolonged intubation defined as continued intubation in the recovery room or ICU/step down unit after surgery,)
  * Nerve injuries due to patient positioning
  * Other intraoperative injuries
* Examples of postoperative adverse events

  * Postoperative bleeding requiring transfusion or reoperation or another procedure
  * Bowel obstruction
  * Anastomotic leak
  * Anastomotic stricture/ stenosis
  * Clostridium difficile infection
  * Liver failure
  * Pancreatitis
  * Peritonitis
  * Acid reflux
  * Stomach or intestine ulceration
  * Wound adverse events: Surgical site Infection-superficial/deep (incisional dehiscence)
  * Deep Venous Thrombosis (DVT)
  * Genitourinary adverse events (Urinary Tract Infection (UTI) requiring antibiotics)
  * Cardiac Adverse events (Atrial arrhythmia requiring treatment, Ventricular arrhythmia requiring treatment, cardiac arrest with CPR, MI)
  * New onset renal failure (per the RIFLE criteria)
  * Sepsis requiring antibiotics
  * Other adverse events: includes any cardiac, pulmonary, gastrointestinal, genitourinary, and neurological adverse events outside of those already listed above

Pre-existing conditions are not reportable as adverse events unless the condition worsens or continues after the procedure. Any events inherent to the procedure are not reportable as adverse events unless the condition worsens or continues after the procedure beyond the expected time frame. Some examples of non-reportable adverse events are listed below:

* Anesthesia related nausea/vomiting occurring <24hrs after surgery
* Leukocytosis as a result of normal post-operative stress response occurring <72hrs after surgery

ELIGIBILITY:
Inclusion Criteria:

* Subject was 18 years or older at the time of procedure
* Subject who has undergone either laparoscopic or robotic-assisted RYGB or SG between the time frame of 30 days prior to institution's IRB approval date and the year 2017
* Subject has one of the below qualifications:

  1. Body mass index (BMI) > 40 kg/m2 or more than 100 pounds overweight OR
  2. BMI > 35 kg/m2 and one of the following obesity-related co-morbidities such as type II diabetes mellitus, hypertension, sleep apnea and other respiratory disorders, non- alcoholic fatty liver disease, osteoarthritis, lipid abnormalities, gastrointestinal disorders, or heart disease.

Exclusion Criteria:

* Subject who underwent RYGB or SG as an emergent procedure
* Subject who underwent RYGB or SG as revisional bariatric procedure
* Subject who underwent RYGB or SG as a secondary (concomitant) procedure and not as a primary procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a multi-center, retrospective chart review study of all consecutive cases of RYGB and SG, performed by participating surgeons at their respective institutions that meet the study inclusion and exclusion criteria.
  The chart review will be performed in a reverse chronological order starting at a minimum of 30 days prior to IRB approval of the study at the site until and going back to 2017 (i.e. most current cases in 2020 and chronologically going back through 2017). Study initiation at the participating site will occur once a research agreement has been executed between Intuitive Surgical and the participating institution/ investigator and after IRB approval has been obtained.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-06-26 (Actual); Primary Completion 2025-04-08 (Estimated); Study Completion 2025-04-08 (Estimated)

PRIMARY OUTCOMES:
Pre-Operative Information: | January 1, 2017 -May 2020
  Collection of Demographics data: gender, age in years Collection of pre-operative medical history: diabetes status, cardiopulmonary disease, hypertension diagnosis, previous abdominal surgery Collection of Demographics patient characteristics: BMI, ASA Class, tobacco use
Intra-Operative Data: | January 1, 2017 -May 2020
  Operative time
Post-Operative Data (up to discharge) | January 1, 2017 -May 2020
  Post-operative data collection such as adverse events, discharge status, hospital length of stay, information on enhanced recovery program
Short-Term Follow-Up Data (up to 30 days post-discharge): | January 1, 2017 -May 2020
  Data collection of events such as Adverse events up to 30 days, re- admissions, re-operations related to the index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Sachin S Kukreja, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Minimally Invasive Surgical Associates, Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No